CLINICAL TRIAL: NCT03054077
Title: Reducing Anxiety in Children Undergoing Procedures
Acronym: REACH-UP!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HM200008056
Record Dates: First submitted 2017-01-31; First posted 2017-02-15 (Actual); Results first posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-09

CONDITIONS: Ambulatory Surgery
Keywords: pre-procedural anxiety; children; pediatric sedation

STUDY DESIGN:
Intervention Model Description: RCT with a control arm equivalent to current standard of care and an intervention arm that includes standard of care plus the addition of an iPad with downloaded games.
Who Masked: Investigator
Masking Description: Blinding occurs through the randomization. Once the assignment to either group 1 (control) or group 2 (intervention) occurs all participants, care providers and investigators will be aware of which group is which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control or Group 1 (No Intervention): This group receives standard of care for the child receiving a sedated procedure. There is no intervention for this group.
- Intervention group or Group 2 (Experimental): This group receives an iPad with downloaded games to play while waiting for the sedation/procedure and then resume play upon return to the recovery area and awakening.
  Interventions: Other: iPad with downloaded games

INTERVENTIONS:
Other: iPad with downloaded games — iPad with downloaded games will be given to children randomized to group 2 for use during their time in the peri-operative unit
  Arms: Intervention group or Group 2

SUMMARY:
This is a small pilot, feasibility study designed as a quality improvement project. The purpose is to identify anxiety in children aged 4-12 years who will receive a sedated procedure and to see if the use of an iPad as a focused activity will decrease the level of anxiety through a small randomized control trial in the Children's Perioperative Unit.

DETAILED DESCRIPTION:
Description: The study is a quality improvement project and designed as a small pilot randomized control trial. Participants will be randomly assigned to either Group 1 (no intervention) or Group 2 (iPad intervention) via a number generator.

Children randomized to Group 1 receive the standard of care with observation and scoring of the mYPAS-SF occurring at three time points (T1 pre-operative holding area-patient room which is private, T2 induction of anesthesia, T3 awakening from sedation post procedure).

Children randomized to Group 2 will be observed at the same time points (T1, T2, T3) but will additionally interact with an iPad that has a selection of 3 games downloaded (3 games for children ages 4-7 and 3 games for children ages 8-12). The iPad is introduced in between T1 and T2 and then resumed at T3 until discharge from the clinical unit.

Process: Following IRB approval, the steps of the study are:

1. . Subjects meeting inclusion criteria (age, first sedated procedure, English speaking) will be identified through daily review of scheduled patient lists by study team members. (CPU Nurse Champions, PI).
2. . Potential subjects will be approached in a private area when they arrive for the procedure to make sure they meet the eligibility criteria. Information concerning the study will be presented by the CPU Nurse Champion, PI or Research Assistant.
3. . If the family is interested in participating in the study, further explanation and consent and assent (as appropriate) will be obtained by the PI or the Research Assistant from the parent and the child.
4. . A demographic questionnaire will be completed following project consenting and enrollment for both groups.
5. . The mYPAS-SF (screening tool that requires a 30 second observation at three distinct time points) will be completed for both groups.
6. . The iPad will be given to participants randomized to Group 2 T1- Child observed in the private holding room area (observation occurs after getting settled in the private room prior to the procedure)

T2-Child observed prior to the induction of anesthesia (observation occurs just prior to the administration of anesthesia).

T3-Child observed upon return to private holding area and awakening from anesthesia (observation occurs when child awakens from the anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* Children admitted for a sedated procedure
* Must be first sedated procedure
* English speaking
* ages 4-12

Exclusion Criteria:

* Non English speaking
* Children younger than 4 and older than 12 years
* Children with developmental disabilities

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Shockey, DNP, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Health System, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No anticipated sharing IPD

REFERENCES:
- [Background] Banchs RJ, Lerman J. Preoperative anxiety management, emergence delirium, and postoperative behavior. Anesthesiol Clin. 2014 Mar;32(1):1-23. doi: 10.1016/j.anclin.2013.10.011. PMID 24491647
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kain ZN, Caldwell-Andrews AA, Mayes LC, Weinberg ME, Wang SM, MacLaren JE, Blount RL. Family-centered preparation for surgery improves perioperative outcomes in children: a randomized controlled trial. Anesthesiology. 2007 Jan;106(1):65-74. doi: 10.1097/00000542-200701000-00013. PMID 17197846

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control or Group 1 | Intervention Group or Group 2
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control or Group 1 | Intervention Group or Group 2 | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Scores With the Addition of the iPad Intervention-Comparing Group 1 to Group 2
Description: The Modified Yale Preoperative Anxiety Scale- Short form (mYPAS-SF) Ratings produce 4 mYPAS scores (1 for each time point)
  Areas scored:
  Activity (1,2,3, or 4) Vocalizations (1,2,3,4,5,or 6) Emotional Expressivity (1,2,3, or 4) State of Apparent arousal (1,2,3, or 4) Scoring: Each score is calculated by dividing each item rating by the highest possible rating (i.e., 6 for the "vocalizations" item and 4 for all other items), adding all the produced values, dividing by 5, and multiplying by 100.
  This calculation produces a score ranging from 23.33 to 100, with higher values indicating higher anxiety.
  Comparison of scores between Group 1 and Group 2 to see if changes in anxiety scores occurred with the addition of the iPad.
  All data will be gathered with review at the close of the study which is anticipated to occur in 5/20/2017.
Time Frame: Immediately following enrollment, immediately before anesthesia, and post-op assessed up to 10 minutes
Population: All participants for whom 3 time points were collected at Baseline T1, T2, and T3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control or Group 1 | Intervention Group or Group 2
Number analyzed (Participants) | 11 | 11
units on a scale
  Time Point 1 | 25 [19.81 to 30.15] | 29.69 [18.73 to 40.65]
  Time Point 2 | 28.82 [19.55 to 38.09] | 24.83 [21.23 to 28.43]
  Time Point 3 | 34.09 [13.19 to 54.99] | 26.56 [15.75 to 37.37]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control or Group 1 | Intervention Group or Group 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT03054077/Prot_SAP_ICF_000.pdf